CLINICAL TRIAL: NCT01193972
Title: Decision Aid Development for Cigarette Smokers Undergoing Surgery: Specific Aim 1
Brief Title: Decision Aid Development for Smokers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: David Warner, MD, Mayo Clinic
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 10-005126
Record Dates: First submitted 2010-08-31; First posted 2010-09-02 (Estimated); Last update posted 2013-02-27 (Estimated); Status verified 2013-02

CONDITIONS: Smoking; Elective Surgery
Keywords: Smoking cessation; Smoking; Tobacco
MeSH Terms: conditions — Smoking; Smoking Cessation | interventions — Decision Support Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Decision aid — Decision aid to assist patients in making a decision about smoking during the perioperative period

SUMMARY:
A decision aid tool will be developed using participatory research approach. The decision aid will be targeted to cigarette smokers scheduled for elective surgery.

ELIGIBILITY:
Inclusion:

* Current cigarette smoker having elective surgery at Mayo Clinic Rochester and is scheduled to be seen at Preoperative Evaluation Center.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2010-09; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Score on Decisional Conflict Scale and COMRADE Scale | Perioperative period

CONTACTS AND LOCATIONS:
Overall Officials: David Warner, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States